CLINICAL TRIAL: NCT00636870
Title: A Randomized, Double-blind, Repeat-dose, Crossover Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Desloratadine (Clarinex®) Compared to Fexofenadine (Allegra®) in Healthy Adults Who Have Been Identified as Slow Metabolizers for Desloratadine.
Brief Title: Fexofenadine (Allegra®) in Healthy Adults Who Have Been Identified as Slow Metabolizers for Desloratadine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M016455_4124
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — fexofenadine

INTERVENTIONS:
Drug: Fexofenadine

SUMMARY:
To evaluate the single-dose and steady-state pharmacokinetics of desloratadine and fexofenadine in desloratadine slow metabolizers. To evaluate the safety and tolerability of desloratadine compared to fexofenadine following single and multiple oral doses administered to desloratadine slow metabolizers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, non-smoking males and females between 18 and 55 years of age, inclusive; Whites of European or North American heritage and Blacks of African or Caribbean heritage.

Exclusion Criteria:

* Any past or present clinically relevant abnormality, medical condition, or circumstance making the subject unsuitable for participation in the study.
* Historical, clinical, or laboratory evidence of liver disease including but not limited to transaminase activity concentrations >2.5 times the upper limit of the reference range.
* Active peptic ulcer disease or a history of gastrointestinal surgery within the last 6 months.
* History of cholecystectomy.
* History of malignancy within the last 5 years (except basal cell carcinoma, which must be in remission for at least 6 months prior to the study.
* Pregnant or lactating females or females of childbearing potential who are unwilling to use reliable, medically accepted methods of contraception. If subjects who are not sexually active with members of the opposite sex become so during the study, these subjects must agree to use a medically accepted method of contraception.
* History of hypersensitivity or intolerability to either desloratadine or fexofenadine or other antihistamines.
* Treatment with other antihistamines in the last month before study entry.
* Use of any prescription or over-the-counter medications or dietary/herbal supplements (with the exception of oral or implanted contraceptives) within 1 week or 5 half-lives, whichever is longer, of the study.
* History of alcoholism or drug abuse within 12 months of the study.
* Ingestion of alcohol within 1 week of the first dose of study medication.
* Ingestion of grapefruit or grapefruit juice within 1 week of the study and a willingness to abstain from the consumption of grapefruit or grapefruit juice for the duration of the study.
* Participation in any other clinical trial or use of an investigational product within 30 days of entry into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2003-02; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Endpoints will be the AUC and Cmax for desloratadine, 3-OH desloratadine, and fexofenadine. | Serial, Trough, and Terminal blood samples over 8 days.

SECONDARY OUTCOMES:
Endpoints will include Tmax, elimination half-life (t1/2), and accumulation index, as the data permit. | Serial, Trough, and Terminal blood samples over 8 days.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States